CLINICAL TRIAL: NCT00239668
Title: Multicenter Benchmarking of Functional and Psychosocial Outcomes of Pediatric Burn Survivors
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Ronald G. Tompkins, Principal Investigator, Massachusetts General Hospital
Other Study IDs: 2001-P-000452/19
Record Dates: First submitted 2005-10-13; First posted 2005-10-17 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2019-03

CONDITIONS: Burn
Keywords: Burns; Functional; Psychosocial; Recovery; Long-term; Pediatric; Surgical; Outcomes; Benchmarking
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to establish an expected recovery trajectory (recovery model) in terms of physical and psychological function of the pediatric burn patient.

DETAILED DESCRIPTION:
The successful advancement of treatment for burns allows us now to save lives of children who sustain massive burn injuries. The purpose of this study is to establish an expected recovery trajectory (recovery model) in terms of the physical and psychological function for pediatric burn patients by assessing prospectively the outcomes of burn children who are treated at the four Shriners Hospitals for Children (SHC) burns hospitals. The study hopes to develop valid benchmarking of outcomes between the four hospitals and therefore, best practices will be utilized. This recovery trajectory will be used as a benchmark for functional and psychosocial outcomes following burn injury.

* Participants in the study complete a series of self reporting questionnaires over a forty-eight month period. There are a total of nine time points during the forty-eight month commitment when questionnaires are given to parent and/or guardian and patients if they are 11 years or older.
* Patients who undergo a reconstructive surgical procedure during their enrollment will fill a set of questionnaires related to the effects of the surgical procedure on their long-term recovery. The surgical procedure is not an intervention because of the study, it is part of their long-term follow-up care after their acute phase. There will be a pre-op and a six and twelve month post-op questionnaire.
* The aim of this study is to develop an expected trajectory recovery model in terms of physical and psychological functioning. Analysis of the data using validated burn specific questionnaires will allow benchmarking of outcomes between the four Shriners Burns Hospitals. We aim to determine predictors of positive outcomes and focus on them as a standard of practice.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric burn patients 18 years or less at time of injuries.
* All high risk patients admitted for burn treatment with injuries >/= 20% total body surface area (tbsa), </= 20% tbsa to critical areas: hands, feet, face, and genitalia.
* All low risk </= 20% to non critical areas.
* Electrical, flame, scald, and chemical burns of at least a second degree nature.
* English and Spanish speaking patients admitted to Shriners Hospital within 30 days of injury

Exclusion Criteria:

* First degree burns
* Patients admitted >30 days post acute injury.
* Patients that speak a language other than English or Spanish.
* Patients who decline to be in the study.
* Patients with a non-burn injury

Ages: 1 Day to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients admitted to Shriners Hospitals-Boston,MA Cincinnati,OH, Galveston,TX and Sacramento, CA burn hospitals with a diagnosis of burn injury.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2000-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G. Tompkins, MD, ScD, Principal Investigator — MGH, Shriners Burn Hospital-Boston
Locations (4):
- United States (4):
  - Shriners Hospital for Children - Sacramento, Sacramento, California
  - Shriners Hospital for Children - Boston, Boston, Massachusetts
  - Shriners Hospital for Children - Cincinnati, Cincinnati, Ohio
  - Shriners Hospital for Children - Galveston, Galveston, Texas

REFERENCES:
- [Derived] Herndon DN, Voigt CD, Capek KD, Wurzer P, Guillory A, Kline A, Andersen CR, Klein GL, Tompkins RG, Suman OE, Finnerty CC, Meyer WJ, Sousse LE. Reversal of Growth Arrest With the Combined Administration of Oxandrolone and Propranolol in Severely Burned Children. Ann Surg. 2016 Sep;264(3):421-8. doi: 10.1097/SLA.0000000000001844. PMID 27433905
- [Derived] Carey K, Kazis LE, Lee AF, Liang MH, Li NC, Hinson MI, Lydon MK, Bauk H, Shapiro GD, Tompkins RG; Multi-Center Benchmarking Study Working Group. Measuring the cost of care for children with acute burn injury. J Trauma Acute Care Surg. 2012 Sep;73(3 Suppl 2):S229-33. doi: 10.1097/TA.0b013e318265c88a. PMID 22929551
- [Derived] Murphy JM, Kazis LE, Li NC, Lee AF, Hinson MI, White GW, Stoddard FJ, Palmieri TL, Meyer WJ 3rd, Liang MH, Tompkins RG; Multi-Center Benchmarking Study Working Group. Test performance characteristics of a case-finding psychosocial questionnaire for children with burn injuries and their families. J Trauma Acute Care Surg. 2012 Sep;73(3 Suppl 2):S221-8. doi: 10.1097/TA.0b013e318265c86b. PMID 22929550
- [Derived] Meyer WJ 3rd, Lee AF, Kazis LE, Li NC, Sheridan RL, Herndon DN, Hinson MI, Stubbs TK, Kagan RJ, Palmieri TL, Tompkins RG; Multi-Center Benchmarking Study Working Group. Adolescent survivors of burn injuries and their parents' perceptions of recovery outcomes: do they agree or disagree? J Trauma Acute Care Surg. 2012 Sep;73(3 Suppl 2):S213-20. doi: 10.1097/TA.0b013e318265c843. PMID 22929549
- [Derived] Palmieri TL, Nelson-Mooney K, Kagan RJ, Stubbs TK, Meyer WJ 3rd, Herndon DN, Hinson MI, Lee AF, Li NC, Kazis LE, Tompkins RG; Multi-Center Benchmarking Study Working Group. Impact of hand burns on health-related quality of life in children younger than 5 years. J Trauma Acute Care Surg. 2012 Sep;73(3 Suppl 2):S197-204. doi: 10.1097/TA.0b013e318265c7ff. PMID 22929547
- [Derived] Warner P, Stubbs TK, Kagan RJ, Herndon DN, Palmieri TL, Kazis LE, Li NC, Lee AF, Meyer WJ 3rd, Tompkins RG; Multi-Center Benchmarking Study Working Group. The effects of facial burns on health outcomes in children aged 5 to 18 years. J Trauma Acute Care Surg. 2012 Sep;73(3 Suppl 2):S189-96. doi: 10.1097/TA.0b013e318265c7df. PMID 22929546
- [Derived] Kazis LE, Lee AF, Hinson M, Liang MH, Rose MW, Palmieri TL, Meyer WJ 3rd, Kagan RJ, Li NC, Tompkins RG; Multi-Center Benchmarking Study Working Group. Methods for assessment of health outcomes in children with burn injury: the Multi-Center Benchmarking Study. J Trauma Acute Care Surg. 2012 Sep;73(3 Suppl 2):S179-88. doi: 10.1097/TA.0b013e318265c552. PMID 22929545
- [Derived] Tompkins RG, Liang MH, Lee AF, Kazis LE; Multi-Center Benchmarking Study Working Group. The American Burn Association/Shriners Hospitals for Children Burn Outcomes Program: a progress report at 15 years. J Trauma Acute Care Surg. 2012 Sep;73(3 Suppl 2):S173-8. doi: 10.1097/TA.0b013e318265c53e. PMID 22929544
- [Derived] Jeschke MG, Gauglitz GG, Kulp GA, Finnerty CC, Williams FN, Kraft R, Suman OE, Mlcak RP, Herndon DN. Long-term persistance of the pathophysiologic response to severe burn injury. PLoS One. 2011;6(7):e21245. doi: 10.1371/journal.pone.0021245. Epub 2011 Jul 18. PMID 21789167